CLINICAL TRIAL: NCT03405454
Title: A Multicentre Phase II Randomised Trial of Durvalumab (MEDI4736) Versus Physician's Choice Chemotherapy in Recurrent Ovarian Clear Cell Adenocarcinomas (MOCCA)
Brief Title: A Multicentre Phase II Trial of Durvalumab Versus Physician's Choice Chemotherapy in Recurrent Ovarian Clear Cell Adenocarcinomas
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GY02/09/16
Record Dates: First submitted 2017-10-19; First posted 2018-01-23 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2018-03

CONDITIONS: Ovarian Clear Cell Carcinoma
MeSH Terms: interventions — durvalumab

STUDY DESIGN:
Intervention Model Description: Patients will be randomized 2:1 to receive either durvalumab at a dose of 1500mg every four weeks for a maximum of 24 months or physician's choice of chemotherapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard chemotherapy (Active Comparator): Patients on physician's choice of chemotherapy are allowed to receive any systemic chemotherapy either as a single agent or in combination. However, biologics( including bevacizumab) and oral tyrosine kinase inhibitors will not be allowed for patients on this arm
  Interventions: Drug: standard chemotherapy
- durvalumab (Experimental): Patients on durvalumab will be given at 1500mg fixed dose every 4 weeks for 24 months
  Interventions: Drug: durvalumab

INTERVENTIONS:
Drug: durvalumab — Durvalumab will be given at 1500mg fixed dose every 4 weeks for 24 months or until the appearance of significant treatment-related toxicity or disease progression
  Arms: durvalumab
Drug: standard chemotherapy — chemotherapy treatment will be administered as per local institutional guidelines
  Arms: standard chemotherapy

SUMMARY:
The purpose of this study is to find out if treatment with a study drug, durvalumab has beneficial effects in people who have recurrent ovarian clear cell cancer and to determine what effects (both good and bad) it has on them and their cancer.

DETAILED DESCRIPTION:
The purpose of this study is to find out if treatment with a study drug, durvalumab has beneficial effects in patients who have recurrent ovarian clear cell cancer and to determine what effects (both good and bad) it has on them and their cancer.

In the recurrent ovarian clear cell cancer (OCCC) setting, responses to further lines of chemotherapy are uniformly low. Given the limited benefit observed from chemotherapy treatments, there is now great interest in the development of molecular targeted therapy for the treatment of OCCC, including immunotherapy.

Researchers have found that sometimes the body's own immune system may be able to slow down or control cancer growth. Sometimes though, this natural immune system response stops, and the cancer cells are not killed by the immune system. Research has shown that in some patients, proteins on the surface of cancer cells and immune cells bind together and send signals that stop the immune cells from killing the cancer cells. One such protein is called Programmed Cell Death Ligand 1 or PD-L1 for short. New drugs like durvalumab work to block this signal and to increase the immune response against cancer cells. Durvalumab is an antibody to PDL1 (a protein that binds to PD1 and blocks the anti tumour activity of immune cells), and it is hoped that by blocking the interaction between PDL1 and PD1, the immune cells will once again be able to attack the cancer cells and thus prevent or slow down cancer growth.

This will be the first study to evaluate the efficacy of durvalumab in patients with recurrent ovarian clear cell carcinomas.

ELIGIBILITY:
Patient Inclusion Criteria

Patients will be eligible for inclusion in this study if all of the following criteria apply:

1. Provision of signed, written and dated informed consent prior to any study specific procedure
2. Female aged 18 years (21 years in Singapore) or older
3. Have histologically documented diagnosis of ovarian clear cell carcinoma as evidenced by WT1 negativity. For tumors with a mixed histology, at least 70% of the tumor must consist of clear cell carcinoma.
4. Provision of an archived tumour tissue block (or at least 10 newly cut unstained slides) where such samples exist in a quantity sufficient to allow for analysis
5. Patients must have had a prior line of platinum-based chemotherap y in the course of their treatment paradigm
6. A maximum of 4 prior lines of systemic treatment regimens will be allowed and may include chemotherapy and biologics (prior immune checkpoint inhibitor treatment will not be permitted).
7. Meet RECIST criteria (version 1.1) within 28 days of start of treatment by having measurable disease defined as one or more lesions that can be accurately measured at baseline as ≥ 10mm in the longest diameter (except lymph nodes which must have a short axis of ≥ 15mm with CT or MRI and which is suitable for repeated measurements). Patients must have radiographic evidence of disease progression following most recent line of treatment. Areas of previous radiation may not serve as measurable disease unless there is evidence of progression post radiation.
8. At time of registration, if the patient has had previous treatment it must have been at least 4 weeks since major surgery or radiation therapy; four weeks from any other previous anti-cancer therapy including biologics. Patients must have recovered from their treatment-related events to ≤1 with the exception of alopecia and neuropathy (≤ 2 sufficient).
9. Have clinically acceptable laboratory screening results within certain limits specified below:

   * AST and ALT ≤ 2.5 times upper limit of normal (ULN), with the exception of:

     i. Patients with documented liver metastasis: AST and/or ALT ≤ 5 X ULN
   * Total bilirubin ≤ ULN; patients with known Gilbert disease who have serum bilirubin level ≤ 3 X ULN may be enrolled
   * Creatinine ≤ 1.5 x UL
   * Absolute neutrophil count ≥ 1500 cells/mm
   * Platelets ≥ 100,000/mm3
   * Hemoglobin ≥ 9.0 g/dl
10. Have an ECOG performance status of ≤ 2.
11. Women of child-producing potential who are sexually active with a non sterilized male partner must agree to use at least one highly effective contraceptive method prior to study entry, during study participation, and for at least 90 days after the last administration of durvalumab
12. A serum pregnancy test within 72 hours prior to the initiation of therapy will be required for women of childbearing potential
13. Have the ability to understand the requirements of the study, provide written informed consent, abide by the study restrictions, and agree to return for the required assessments.
14. Life expectancy greater than 12 weeks

Patient Exclusion Criteria

Patients will not be eligible for inclusion in this study if any of the following criteria apply:

1. Women who are pregnant or nursing
2. Prior exposure to an immune checkpoint inhibitor (anti-PD-1 or anti-PDL-1 antibody)
3. Any prior Grade ≥3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent, or any unresolved irAE >Grade 1
4. Active or prior documented autoimmune disease within the past 2 years. NOTE: Patients with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded.
5. Active or prior documented inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis)
6. Have active, acute, or chronic clinically significant infections or bleeding including but not limited to active bleeding diatheses, patients known to have evidence of acute or chronic hepatitis B, hepatitis C or human immunodeficiency virus (HIV),
7. History of primary immunodeficiency
8. History of allogeneic organ transplant
9. Known history of previous clinical diagnosis of tuberculosis
10. Have uncontrolled hypertension (systolic blood pressure greater than 150mmHg or diastolic blood pressure greater than 100mmHg);
11. Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or greater), myocardial infarction within the previous 3 months or unstable angina
12. Chronic atrial fibrillation or QTc interval corrected for heart rate of greater than 470 msec. calculated from 3 electrocardiograms (ECGs) using Frediricia's Correction.

    • By Fridericia's formula: QTc = QT/(RR^0.33) Where - RR interval = 60 / HR ; HR = Heart rate in beats per minute.
13. Have additional uncontrolled serious medical or psychiatric illness.
14. Recent major surgery within 4 weeks prior to entry into the study (excluding the placement of vascular access) that would prevent administration of investigational product
15. Require therapeutic doses of anti-coagulation with warfarin or warfarin derivatives. However, treatment with low molecular weight heparin (LMWH) is allowed.
16. Brain metastases or spinal cord compression unless asymptomatic, treated and stable off steroids and anti-convulsants for at least 1 month prior to entry into the study
17. History of leptomeningeal carcinomatosis
18. History of another primary malignancy unless treated with curative intent and with no known active disease ≥5 years except:

    * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
    * Adequately treated carcinoma in situ without evidence of disease eg, cervical cancer in situ
19. Absence of a tumour sample (archival and/or recent).
20. Current or prior use of systemic immunosuppressive medications within 28 days before the first dose of durvalumab (including but not limited to prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents)

    * Patients on systemic corticosteroids at physiological doses, which do not exceed 10 mg/day of prednisone, or an equivalent corticosteroid are allowed
    * The use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) is allowed.
21. Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving durvalumab
22. Patients who are pregnant, breast-feeding or of reproductive potential who are not employing an effective method of birth control
23. Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results

Ages: 21 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only the females are affected by the ovarian clear cell carcinoma (OCCC).
Enrollment: 46 (Estimated)
Dates: Start 2017-10-09 (Actual); Primary Completion 2021-09-15 (Estimated); Study Completion 2022-03-15 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 4 years
  Progression free survival (PFS) is defined as the time from the first day of treatment to the first observation of radiological or clinical disease progression or death due to any cause or last follow-up. The progression will be defined by RECIST criteria v1.1 for patients on the chemotherapy arm which includes first instance of more than 20% increase in the sum of diameters or unequivocal progression in non-target disease. The sum of the diameters (longest for non-nodal lesions, short axis for nodal lesions) is calculated at baseline and at each tumor assessment.

SECONDARY OUTCOMES:
Objective Response Rate | 4 years
  Objective response rate (ORR) is defined as the percentage of subjects with a confirmed CR or PR as per RECIST 1.1 criteria. Response will be evaluated every 8 weeks while on treatment.
Overall survival | 4 years
  Overall survival (OS) is measured as time from the first day of treatment to the time of death from any cause.
Health related Quality of life (HRQOL) | 4 years
  HRQOL will be measured using European Organization for Research and Treatment of Cancer Core questionnaire.
Adverse event profile | 4 years
  Adverse event profile of durvalumab in this patient population as measured by CTCAE 4.0 criteria

CONTACTS AND LOCATIONS:
Overall Officials: David SP Tan, Principal Investigator — National University Hospital, Singapore
Locations (2):
- Singapore (2):
  - National University Hospital, Singapore
  - National Cancer Centre, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mackay HJ, Brady MF, Oza AM, Reuss A, Pujade-Lauraine E, Swart AM, Siddiqui N, Colombo N, Bookman MA, Pfisterer J, du Bois A; Gynecologic Cancer InterGroup. Prognostic relevance of uncommon ovarian histology in women with stage III/IV epithelial ovarian cancer. Int J Gynecol Cancer. 2010 Aug;20(6):945-52. doi: 10.1111/IGC.0b013e3181dd0110. PMID 20683400
- [Background] Kobel M, Kalloger SE, Huntsman DG, Santos JL, Swenerton KD, Seidman JD, Gilks CB; Cheryl Brown Ovarian Cancer Outcomes Unit of the British Columbia Cancer Agency, Vancouver BC. Differences in tumor type in low-stage versus high-stage ovarian carcinomas. Int J Gynecol Pathol. 2010 May;29(3):203-11. doi: 10.1097/PGP.0b013e3181c042b6. PMID 20407318
- [Background] Yamagami W, Aoki D. Annual report of the Committee on Gynecologic Oncology, the Japan Society of Obstetrics and Gynecology. J Obstet Gynaecol Res. 2015 Feb;41(2):167-77. doi: 10.1111/jog.12596. Epub 2014 Nov 5. PMID 25370711
- [Derived] Ngoi NY, Heong V, Ow S, Chay WY, Kim HS, Choi CH, Goss G, Goh JC, Tai BC, Lim DG, Kaliaperumal N, Au VB, Connolly JE, Kim JW, Friedlander M, Kim K, Tan DS. A multicenter phase II randomized trial of durvalumab (MEDI-4736) versus physician's choice chemotherapy in recurrent ovarian clear cell adenocarcinoma (MOCCA). Int J Gynecol Cancer. 2020 Aug;30(8):1239-1242. doi: 10.1136/ijgc-2020-001604. Epub 2020 Jun 25. PMID 32591370